CLINICAL TRIAL: NCT05543993
Title: Serological and Functional Impact of COVID-19 Vaccination on the Maternal Fetal Unit and Infant Immunity
Brief Title: COVID Booster in Pregnancy and Lactation
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Nemours Childrens Health (Unknown)
Responsible Party: Principal Investigator, Rupsa C. Boelig, Assistant Professor, Thomas Jefferson University
Other Study IDs: 22F.452
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: vaccine; COVID-19 vaccine; booster; pregnancy; breastfeeding; immunity
MeSH Terms: conditions — COVID-19; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood Cord blood Breastmilk Infant blood Infant oral
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- COVID-19 booster in pregnancy: Pregnant singletons who have received COVID-19 booster in pregnancy
  Interventions: Drug: Bivalent COVID-19 Booster
- COVID-19 booster in breastfeeding: Breastfeeding individuals who have received COVID-19 booster while breastfeeding
  Interventions: Drug: Bivalent COVID-19 Booster

INTERVENTIONS:
Drug: Bivalent COVID-19 Booster — Bivalent COVID-19 Booster by Pfizer or Moderna

SUMMARY:
This is a prospective longitudinal cohort study to evaluate the impact of COVID-19 vaccination and booster on maternal and infant immunity against COVID-19 variants over time.

DETAILED DESCRIPTION:
We will enroll 100 pregnant patients who have received COVID-19 mRNA booster as well as 100 breastfeeding patients who have received COVID-19 mRNA booster. Participants will be following longitudinally through 3 months post partum, or 3 months post enrollment for those in the breastfeeding cohort. Maternal blood will be collected, as will cordblood at delivery, breastmilk, and infant samples.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Received mRNA bivalent COVID-19 booster during 1) pregnancy or 2) breastfeeding

Exclusion Criteria:

* Multifetal gestation
* Unable to provide consent

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Pregnant singleton gestation who have received bivalent COVID-19 mRNA booster in pregnancy
  2. Breastfeeding individuals who have recieved bivalent COVID-19 mRNA booster
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Maternal Serological Profile | 3 months
  Quantitative Maternal IgG to SARS CoV2 spike and other domains
Maternal Functional Immunity | 3 months
  Quantitative Antibody neutralization capacity

SECONDARY OUTCOMES:
Infant serological profile | 3 months old
  Quantitative IgG to SARS CoV2
Infant functional immunity | 3 months old
  Quantitative Antibody neutralization capacity
Breastmilk serological profile | 3 months
  Quantitative IgA to SARS CoV2
Infant oral immunity | 3 months
  Quantitative Salivary SARS CoV2 IgG

CONTACTS AND LOCATIONS:
Overall Officials: Rupsa C Boelig, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected will be shared in a de-identified manner upon completion of appropriate data sharing agreements
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 12 months after publication of primary results and for up to 2 years
Access Criteria: Data collected will be shared in a de-identified manner upon completion of appropriate data sharing agreements